CLINICAL TRIAL: NCT06235398
Title: Upfront Related Donor Transplantation in Patients With Myelodisplatic Syndrome : a Phase 2 Trial
Acronym: FIRST ALLO MDS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP221273
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-08

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with Myelodysplasic Syndrome diagnosis (Experimental): Adults (Age ≥ 50 and ≤ 70 years) patients with MDS diagnosis for whom transplantation is indicated from a related donor identified.
  Interventions: Biological: Hematopoietic stem-cell transplantation

INTERVENTIONS:
Biological: Hematopoietic stem-cell transplantation — Upfront related donor transplantation

SUMMARY:
Three recent prospective "transplant/no transplant" studies concluded to an advantage of OS with transplantation in patients with high or intermediate-2 IPSS risk (not significant in Kröger's study). No prospective randomized trial has assessed the pre-transplant therapy in MDS patients yet but some information can be extracted from these 3 recent studies. In the French study (n=162), 72% patients with a donor received HSCT, previously treated by hypomethylating agent (HMA) in 71% of them. There was a trend to a better survival in patients achieving a complete remission with pre-graft therapy (HR: 0.55, p=0.088) and higher risk of death in unresponsiveness patients transformed into AML (HR: 2.36, p=0.008). In Nakamura's study (n=384), 83% of patients with a donor were transplanted, previously treated by HMA in 68%2. The multivariable Cox model for Overall Survival (OS) and Leukemia-free survival showed an excess risk in patients treated by HMA. Moreover, responders still have a higher risk of mortality as compared to patients who did not receive any pre-graft therapy (HR: 2.417, p=0.0054). In the German study, the aim was to initiate azacytidine at inclusion and to transplant patients after 4 cycles if a donor was identified1. Among 170 registered patients, 162 initiated 5-aza but 36% of them were "lost during this pre-graft therapy" before allocation to "donor" or "no-donor" arm, for different reasons including death (n=12). After 4 cycles of 5-aza, 79/81 patients "donor arm" were transplanted. The multivariable analysis showed remission status did not influence OS. Those 3 previous clinical trials thus suggest that a substantial number of patients planned for transplantation are not transplanted nowadays while no evidence of HMA benefit before HSCT has been clearly identified. This phase 2 study aim to assess the feasibility of upfront HSCT in patients with high risk MDS in order to increase the probability to be transplanted and to achieve a subsequent remission and better survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 and ≤ 70 years
* An HLA (Human Leukocyte Antigen) matched sibling donor or familial haplo-identical donor has been identified
* The disease fulfills at least one of the following criteria:

  * Intermediate-2 or high risk according to classical International Prognostic Scoring System (IPSS)
  * Intermediate-1 risk if marrow fibrosis > grade I or poor risk cytogenetics according to R IPSS or classified high or very high risk according to Revised International Prognostic Scoring System (R IPSS) or if the MDS is therapy-related neoplasm
* Usual criteria for Hematopoietic Stem Cell Transplantation (HSCT):

  * Eastern Cooperative Oncology Group Score (ECOG) ≤ 2
  * No severe and uncontrolled infection
  * Cardiac function compatible with high dose of cyclophosphamide Left Ventricular Function (LVF) > 50%
  * Adequate organ function: ASAT and ALAT ≤ 2.5N, total bilirubin ≤ 2N, creatinine clearance ≥ 30 ml/min (according to Cockroft formula)
* In case of transplantation with a haploidentical donor, absence of donor specific antibody (DSA) detected in the patient with a MFI >1000 (antibodies directed towards the distinct haplotype between donor and recipient)
* Contraception methods must be prescribed for women of childbearing age during all the study. If cyclophosphamide is used, effective contraceptive methods for men during all their participation in the study
* With health insurance coverage
* With a written informed consent signed

Exclusion Criteria:

* Marrow blast > 15% at time of inclusion
* MDS with excess blast >10% and NPM1 mutation or a recurrent genetic abnormality related to Acute Myeloid Leukemia (AML) (WHO 2022)
* Chemotherapy (AML like intensive chemotherapy or demethylating agent) to treat MDS at the current stage
* Disponibility of an unrelated donor 10/10 (MUD) in absence of geno-identical donor
* Patient with uncontrolled infection
* Cancer in the last 5 years (except basal cell carcinoma of the skin or "in situ" carcinoma of the cervix
* Renal failure with creatinine clearance <30ml / min (according to Cockroft formula)
* With contraindications to treatments used during the research
* Uncontrolled coronary insufficiency, recent myocardial infarction <6 month, current manifestations of heart failure, uncontrolled cardiac rhythm disorders, ventricular ejection fraction <50%
* With heart failure according to NYHA (II or more)
* Patient with seropositivity for HIV or HTLV-1 or active hepatitis B or C defined by a positive PCR Hepatitis B Virus or Hepatitis C Virus
* Yellow fever vaccine or any alive vaccine within 2 months before transplantation
* Pregnancy (β-HCG positive) or breast-feeding
* Who have any debilitating medical or psychiatric illness, which would preclude giving well understand informed consent or optimal treatment and follow-up
* Under protection by law (tutorship or curatorship)

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years after transplantation

SECONDARY OUTCOMES:
Overall survival | 2 years after transplantation
Non-relapse mortality | 2 years after transplantation
Cumulative incidence of transformation into acute myeloid leukemia from inclusion | 2 years after inclusion
Incidence of acute Graft versus Host Disease (GvHD) and grading | 100 days after transplantation
Incidence of chronic GvHD and grading | 2 years after transplantation
Percentage of engraftment | 3 months after transplantation
  Engraftment is defined by hematological recovery and donor chimerism > 95%
Percentage of graft failure | 2 years after transplantation
  Graft failure is defined by acute or late rejection and non-engraftment
Incidence of severe infections | 3 months after transplantation
  Severe infections are defined by Common Terminology of Adverse Events (CTAE) grade 3-4
Incidence of severe infections | 6 months after transplantation
  Severe infections are defined by Common Terminology of Adverse Events grade 3-4
Incidence of severe infections | 12 months after transplantation
  Severe infections are defined by Common Terminology of Adverse Events grade 3-4
Incidence of severe infections | 24 months after transplantation
  Severe infections are defined by Common Terminology of Adverse Events grade 3-4
Incidence of cardiac events | 1 month after transplantation
  CTAE grade 2-4
Incidence of cardiac events | 3 months after transplantation
  CTAE grade 2-4

IPD SHARING:
Plan to Share IPD: Undecided